CLINICAL TRIAL: NCT04033276
Title: A Randomized, Open, Controlled Trial of High Dose IVIG/Rituximab Versus Rituximab in Kidney Transplant Patients With de Novo Donor-specific Antibodies
Brief Title: IVIG/Rituximab vs Rituximab in Kidney Transplant With de Novo Donor-specific Antibodies
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Severance Hospital (Other); GC Biopharma Corp (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20180138795
Record Dates: First submitted 2019-07-24; First posted 2019-07-26 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-05

CONDITIONS: Renal Transplant
MeSH Terms: interventions — Rituximab; Immunoglobulins, Intravenous

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Rituximab (Active Comparator): Inj Rituximab 375mg/m2 IV given on day 0
  Interventions: Drug: Rituximab
- Combination of high-dose IVIG and Rituximab (Active Comparator): IV Rituximab 375mg/m2 on day 0 and IV high-dose IVIG 2g/kg on day 0
  Interventions: Drug: Rituximab; Drug: intravenous immune globulin

INTERVENTIONS:
Drug: Rituximab — IV rituximab
  Other Names: mabthera
Drug: intravenous immune globulin — iv intravenous immune globulin
  Other Names: IVIG-SN
  Arms: Combination of high-dose IVIG and Rituximab

SUMMARY:
The objective of this study was to compare two strategies of de novo donor specific antibodies (DSA) and antibody-mediated rejection (AMR) prevention in renal transplant recipients: high dose intravenous immunoglobulin (IVIG)/rituximab regimens versus rituximab alone.

DETAILED DESCRIPTION:
Although recent advances in immunosuppressive regimens after kidney transplantation (KT) have reduced the incidence and consequences of T-cell-mediated rejection (TCMR) and have improved short-term outcomes, long-term allograft loss attributable to AMR is still responsible for substantial medical and socioeconomic burdens in kidney transplant recipients. Numerous studies have shown that de novo DSA after KT are associated with AMR, which leads to allograft loss. IVIG is a medication that has emerged as a useful tool in modulating immunity, treatment of AMR and in desensitization protocol. Treatment with rituximab or combination of IVIG/rituximab has sought to further diminish antibody production (de novo DSA) in the treatment of AMR. Several studies have been reported, but in the absence of control groups or standardization of treatment, their efficacy is difficult to assess.

ELIGIBILITY:
Inclusion Criteria:

All patients have de novo production of DR or DQ DSA after renal transplantation Inclusion criteria requires all of the following

1. age ≥ 19 years
2. Renal transplants with eGFR ≥ 20 ml/min (by CKD-EPI equation) and change in the eGFR ≤ 20 within 3 months
3. No history of biopsy proven acute T cell mediated rejection or antibody-mediated rejection within 3 months
4. peak MFI of de novo DSA (DR or DQ) ≥ 1000
5. A patient who agree to write a written consent form

Exclusion Criteria:

1. age ≤ 18 years
2. multi-organ transplantation
3. Patients with no history of tacrolimus as immunosuppressants
4. history of allergic or anaphylactic reaction to rituximab
5. human immunodeficiency virus infection
6. active infection
7. pregnancy or lactation
8. history of drug abuse or alcohol abuse within 6 months
9. history of malignancy within 5 years
10. history of treatment for psychiatric problems
11. hematologic or biochemical abnormalities (Hb < 7g/dL, Platelet < 1x105/mm3, AST/ALT > 80IU)
12. A patient who do not want to participate in this study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-01-08 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-05-03 (Actual)

PRIMARY OUTCOMES:
change in delta DSA MFI sum | baseline and 3 months post-treatment, 1 year post-treatment
  change of pre- and post-treatment DSA MFI sum, monitoring DSA during follow-up period

SECONDARY OUTCOMES:
Change in estimated glomerular filtration rate(eGFR) by CKD-EPI equation | baseline and 3 months post-treatment, 1 year post-treatment
  change of pre- and post-treatment eGFR by CKD-EPI equation, monitoring eGFR during follow-up period
Development of antibody-mediated rejection (AMR) | up to 1 year post-treatment
  To identify the development of AMR after treatment during follow-up period

CONTACTS AND LOCATIONS:
Overall Officials: Jaeseok Yang, M.D., Ph.D., Principal Investigator — Seoul National University Hospital
Locations (2):
- South Korea (2):
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim HW, Lee J, Heo SJ, Kim BS, Huh KH, Yang J. Comparison of high-dose IVIG and rituximab versus rituximab as a preemptive therapy for de novo donor-specific antibodies in kidney transplant patients. Sci Rep. 2023 May 11;13(1):7682. doi: 10.1038/s41598-023-34804-6. PMID 37169835